CLINICAL TRIAL: NCT04047888
Title: Assessment of Risk Factors for Childhood Obesity and the Impact of a Nutrition-based Educational Intervention on Infant Feeding, Growth and Body Composition
Brief Title: Assessment of Risk Factors for Childhood Obesity and Nutrition Education Intervention on Infant Growth and Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: EC115-17/18
Record Dates: First submitted 2019-06-15; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-02

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The first sample will be the baseline sample. After that a dose of deuterium oxide will be administered and then two other samples of saliva will be taken at 3 hours and four hour intervals. when the dose has equilibrated with total body water. Saliva samples will be collected using a dry cotton wool swab. With assistance, the swab will be moved around the mouth until the cotton wool is sodden. After removing the plunger from a 20 ml syringe barrel, the cotton wool from the swab will be removed and placed in the barrel of the syringe the plunger will be replaced and used to squeeze the saliva into a cryovial for storage at - 20 degrees centigrade for later analysis of deuterium enrichment by FTIR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Mothers and children in this group will have measurements, questionnaire administration. The children will have routine child care at their health center and mothers will have a 60 minute nutrition-based and non-nutrition based educational message
  Interventions: Other: Nutrition-based education on infant feeding and practices as well as Non nutrition-based educational message
- Control Group: Mothers and babies will have measurements and questionnaire administration and children will receive routine child care at their health centers. These mothers will receive a non-nutrition based educational message only.
  Interventions: Other: Non nutrition-based educational message

INTERVENTIONS:
Other: Nutrition-based education on infant feeding and practices as well as Non nutrition-based educational message — 60 minute educational message at each visit
  Groups: Intervention Group
Other: Non nutrition-based educational message — No nutrition-based education on infant feeding and practices
  Groups: Control Group

SUMMARY:
The period from conception to 2 years of age ('first 1000 days') has been recognized as a critical period for long-lasting programming effects on later obesity and associated NCD and a window of opportunity to implement intervention for reducing and treating childhood obesity. However, there is a dearth of prospective intervention studies that address this nutritional problem in Jamaica and there are no reports of sustainable intervention.

Jamaica is a middle income country in which overweight and obesity in children are also increasing at an alarming rate. The investigators in Jamaica are seeking to provide a more comprehensive knowledge on the link between early life nutrition and later childhood health and to assess the impact of an intervention of infant feeding counselling/education in mothers on growth and body composition in their offspring.

DETAILED DESCRIPTION:
At least 41 million children younger than 5 years are overweight or obese most of whom reside in low-income and middle-income countries (LMIC). Obese children tend to remain obese in adulthood predisposing to the huge personal health and economic burden of the non-communicable diseases (NCD).

Several early life factors identified to contribute to development of obesity and adverse metabolic profile; pre-pregnancy underweight and overweight, high weight gain in early pregnancy in addition to inappropriate infant feeding pattern and rapid weight gain in early life have major role.

The aims of the study are:1) to assess intrauterine and postnatal risk factors for childhood obesity in children followed from the second trimester in mother's pregnancy to age 1 year and 2) to assess the impact of a nutrition-based educational intervention on infant feeding, growth and body composition in the first year of life.

This study design is a cluster randomized clinical trial with key outputs being : 1) The use of deuterium dilution method to provide new data on body composition of mothers from during pregnancy and during infancy in addition to obtain accurate measurement of breastmilk intake 2) new data on the relationship between maternal body composition and/or infant body composition and non-communicable disease risk factors; 3) new data on the impact of a nutrition-based educational on infant's growth and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Women (18-40 years)
* Women 30 -32 weeks gestation
* First or second pregnancy
* Healthy term infants ( > 37 completed weeks)
* Infants with birthweight >2.5kg)

Exclusion Criteria:

* Pre-gestational diabetes
* Pre-gestational hypertension
* Sickle cell disease
* HIV infection,
* Psychiatric disorder
* Gestational diabetes
* Infants with congenital abnormalities
* Infants with chromosomal disorders
* Infants admitted in neonatal period > 48 hours

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will be conducted on Mothers and their babies
Study Population: The target populations from which participants will be selected will consist of pregnant women attending antenatal visits at Public Health Centers in Kingston and St. Andrew (KSA). Mothers will be recruited prior to 30-32 weeks gestation and study measurements will be made in the middle of the third trimesters
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Feeding Questionnaire - first assessment | 2 weeks old
  This questionnaire will describe breastfeeding and complementary feeding practices. Proportions will be used to compare responses between the intervention and control groups. A scale will not be used.
Feeding Questionnaire - second assessment | 4 weeks old
  This questionnaire will describe breastfeeding and complementary feeding practices. Proportions will be used to compare responses between the intervention and control groups. A scale will not be used.
Feeding Questionnaire - third assessment | 3 months old
  This questionnaire will describe breastfeeding and complementary feeding practices. Proportions will be used to compare responses between the intervention and control groups. A scale will not be used.
Feeding Questionnaire - fourth assessment | 6 months old
  This questionnaire will describe breastfeeding and complementary feeding practices. Proportions will be used to compare responses between the intervention and control groups. A scale will not be used.
Feeding Questionnaire - fifth assessment | 12 months old
  This questionnaire will describe breastfeeding and complementary feeding practices. Proportions will be used to compare responses between the intervention and control groups. A scale will not be used.
Child's lean mass and fat mass (body composition) determined using skin fold measurements - first assessment | 6 months old
  Child's fat mass and lean mass (body composition) determined using skin fold callipers
Child's fat mass and lean mass (body composition) determined using Bioelectrical Impedance Analysis (BIA) - first assessment | 6 months old
  Child's fat mass and lean mass (body composition) determined using a Bioelectrical Impedance Analyzer
Child's mid-upper arm circumference - first assessment | 6 months
  Child's mid-upper arm circumference measured using a tape measure
Child's lean mass and fat mass (body composition) determined using skin fold measurements - second assessment | 12 months old
  Child's fat mass and lean mass (body composition) determined using skin fold callipers
Child's fat mass and lean mass (body composition) determined using Bioelectrical Impedance Analysis (BIA) - second assessment | 12 months old
  Child's fat mass and lean mass (body composition) determined using a Bioelectrical Impedance Analyzer
Child's mid-upper arm circumference - second assessment | 12 months old
  Child's mid-upper arm circumference measured using a tape measure
Child's fat mass and lean mass (body composition) determined using deuterium dilution method - first assessment | 6 months old
  Measurement of fat mass and lean mass (body composition) using the deuterium dilution method
Child's fat mass and lean mass (body composition) determined using deuterium dilution method - second assessment | 12 months old
  Measurement of fat mass and lean mass (body composition) using the deuterium dilution method
Child's weight in kilograms - first assessment | 4 weeks old
  Child's weight measured using a digital scale
Child's weight in kilograms - second assessment | 3 months old
  Child's weight measured using a digital scale
Child's weight in kilograms - third assessment | 6 months old
  Child's weight measured using a digital scale
Child's weight in kilograms - fourth assessment | 12 months old
  Child's weight measured using a digital scale
Child's length in centimeters - first assessment | 4 weeks old
  Child's length measured using a stadiometer
Child's length in centimeters - second assessment | 3 months old
  Child's length measured using a stadiometer
Child's length in centimeters - third assessment | 6 months old
  Child's length measured using a stadiometer
Child's length in centimeters - fourth assessment | 12 months old
  Child's length measured using a stadiometer
Child's fat mass and lean mass (body composition) determined using Dual-energy X-ray absorptiometry (DEXA) | 12 months old
  A whole body DEXA scan will be done as described by the International Atomic Energy Agency. A scan takes about 7 minutes.
Child's fat mass and lean mass (body composition) determined using Air Displacement Plethysmography - first assessment | 4 weeks old
  Measurement of child's fat mass and lean mass (body composition) using the Air Displacement Plethysmography
Child's fat mass and lean mass (body composition) determined using the Air Displacement Plethysmography - second assessment | 3 months old
  Measurement of child's fat mass and lean mass (body composition) using the Air Displacement Plethysmography
Child's fat mass and lean mass (body composition) determined using the Air Displacement Plethysmography - third assessment | 6 months old
  Measurement of child's fat mass and lean mass (body composition) using the Air Displacement Plethysmography

SECONDARY OUTCOMES:
Screen time / sleep time questionnaire - first assessment | 3 months old
  This will describe total duration of sleep time and screen viewing time. Child's feeding pattern during the night will also be assessed (if the child fed or did not feed). Proportions will be used to compare responses between the intervention and control groups. Absolute values will also be compared for some questions. A scale will not be used.
Screen time / sleep time questionnaire - second assessment | 6 months old
  This will describe total duration of sleep time and screen viewing time. Child's feeding pattern during the night will also be assessed (if the child fed or did not feed). Proportions will be used to compare responses between the intervention and control groups. Absolute values will also be compared for some questions. A scale will not be used.
Screen time / sleep time questionnaire - third assessment | 12 months old
  This will describe total duration of sleep time and screen viewing time. Child's feeding pattern during the night will also be assessed (if the child fed or did not feed). Proportions will be used to compare responses between the intervention and control groups. Absolute values will also be compared for some questions. A scale will not be used.
Breastmilk intake in child | 3 months old
  To determine the amount of breastmilk consumed. The mother will consume a carefully weighed dose of deuterium. Saliva samples will be collected from the mother and her infant at baseline and at 2 timepoints between 1 and 14 days following dose consumption. Deuterium enrichment will be measured by Fourier transform infrared (FTIR) Spectrometry.
Mother's fat mass and lean mass (body composition) determined using deuterium (2H) dilution technique - first assessment | 30-32 weeks gestation
  Fat mass and lean mass (body composition)determined using deuterium (2H) dilution technique
Mother's fat mass and lean mass (body composition) determined using skin fold measurements - first assessment | 30-32 weeks gestation
  Fat mass and lean mass (body composition) measured using skin fold callipers
Mother's fat mass and lean mass (body composition) determined using Bioelectrical Impedance Analysis (BIA) - first assessment | 30-32 weeks gestation
  Fat mass and lean mass (body composition) measured using BIA analyzer
Mother's weight - first assessment | 30-32 weeks gestation
  Mother's weight measured using a digital scale
Mother's height | 30-32 weeks gestation
  Mother's height measured using a stadiometer
Mother's mid-upper arm circumference - first assessment | 30-32 weeks gestation
  Mother's mid-upper arm circumference measured using a tape measure
Mother's fat mass and lean mass (body composition) determined using skin fold measurements - second assessment | 3 months post natally
  Mother's fat mass and lean mass (body composition) determined using skin fold calliper
Mother's fat mass and lean mass (body composition) determined using Bioelectrical Impedance Analysis (BIA) - second assessment | 3 months post natally
  Fat mass and lean mass (body composition) determined measured using BIA analyzer
Mother's fat mass and lean mass (body composition) using deuterium dilution - second assessment | 3 months post natally
  Fat mass and lean mass (body composition) determined using deuterium dilution during breastmilk assessment
mother's weight - second assessment | 3 months post natally
  mothers weight measured using a scale
mother's mid-upper arm circumference - second assessment | 3 months post natally
  mother's mid-upper arm circumference measured using a tape measure
Mother's fat mass and lean mass (body composition) determined using skin fold measurements - third assessment | 12 months post natally
  Mother's fat mass and lean mass (body composition) determined using skin fold callipers
Mother's fat mss and lean mass (body composition) determined using Bioelectrical Impedance Analysis (BIA) - third assessment | 12 months post natally
  mother's fat mass and lean mass (body composition) determined using BIA analyzer
mother's weight - third assessment | 12 months post natally
  mothers weight measured using a scale
mother's mid-upper arm circumference - third assessment | 12 months post natally
  mother's mid-upper arm circumference measured using a tape measure

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn R Taylor Bryan, PhD, Principal Investigator — University of the West Indies, Mona
Locations (1):
- Tropical Metabolism Research Unit, TMRU University of the West Indies,, Mona, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided